CLINICAL TRIAL: NCT00821522
Title: The Influence of Remote Ischemic Preconditioning on Acute Kidney Injury After Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Kramer, MD (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Robert Kramer, MD, Thoracic Surgery, MD, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3401
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Acute Kidney Insufficiency; Acute Renal Insufficiency; Acute Kidney Injury; Ischemic Preconditioning
Keywords: Acute Kidney Insufficiency; Acute Renal Insufficiency; Acute Kidney Injury; Cardiac Surgical Procedures; Ischemic Preconditioning
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preconditioning (Active Comparator)
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control (No Intervention): Standard clinical management during cardiac surgery.

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Three 5-minute intervals of leg ischemia induced by tourniquet inflation, prior to initiation of cardiopulmonary bypass.
  Arms: Preconditioning

SUMMARY:
Acute kidney injury is associated with cardiopulmonary bypass during heart surgery and its pathogenesis is similar to that of ischemia-reperfusion injury. Remote ischemic preconditioning attenuates myocardial ischemia-reperfusion injury in patients undergoing coronary bypass surgery. The investigators hypothesize that such preconditioning reduces the incidence of acute kidney injury associated with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing heart surgery on cardiopulmonary bypass.

Exclusion Criteria:

* Known peripheral vascular disease of the lower extremities associated with active skin necrosis or infection.
* End-stage renal disease.
* Inability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury, after surgery, as defined by elevation in serum creatinine greater than or equal to 0.3 mg/dl. | 48 hours after surgery.

SECONDARY OUTCOMES:
Oliguria. | 12 hours after surgery.
Incidence of acute kidney injury as defined by post-operative elevation in NGAL. | 3 hours after cardiopulmonary bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Zimmerman, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States